CLINICAL TRIAL: NCT03440931
Title: Monitoring Ovarian Cysts in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 239020
Record Dates: First submitted 2018-01-12; First posted 2018-02-22 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Ovarian Cysts
MeSH Terms: conditions — Ovarian Cysts | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound scan — Transvaginal ultrasound scan to assess ovaries

SUMMARY:
This prospective study will primarily aim to determine what monitoring is required of ovarian cysts when they are diagnosed in pregnancy, as well as what intervention, if any, is necessary. It also aims to identify the prevalence of ovarian cysts in pregnancy and the nature of these cysts, as well as their natural history throughout pregnancy.

DETAILED DESCRIPTION:
The Royal College of Obstetricians and Gynaecologists currently publish guidelines for the management of ovarian cysts in both pre and post-menopausal women. The guidelines for pre-menopausal women do not specifically include pregnant women, and it is known from previous research that the characteristics of ovarian cysts can differ in pregnancy, and therefore appear different on ultrasound scan. Also, where intervention is needed, it is usually surgical which can have high risk implications in pregnancy.

The study will be conducted in the Early Pregnancy and Acute Gynaecology Unit at St. Thomas' Hospital. Any woman who presents with symptoms in early pregnancy (less than 18 weeks) is offered a transvaginal ultrasound scan. If, on this scan, they are found to have an ovarian cyst, they will be considered for the study. Once the ovarian cyst has initially been diagnosed, a confirmatory scan will be carried out by one of the investigators (ie. a clinical fellow, consultant gynaecologist or senior sonographer).

If the cyst is benign in nature and not the cause of acute symptoms, three more transvaginal scans will be carried out by one of the investigators at approximately 12 weeks and 20 weeks (in line with the nuchal translucency scan and anomaly scan), then at 6 weeks post partum. It is intended that all these patients will be managed without surgical intervention.

If there are concerns that the cyst is malignant, the participant would be investigated via the already established pathways. If the participant is at any point in acute pain and the cyst is thought to be the cause of this eg. ovarian torsion or cyst rupture, then a clinical decision would be made regarding surgical intervention.

The total study period will be up to 16 months. This includes a 6 month recruitment period, then following up each participant until 6 weeks post delivery.

ELIGIBILITY:
Inclusion Criteria:

- Age 16-50 Pregnant Scanned in the Early Pregnancy Unit at St. Thomas' Hospital (either as a walk in patient / a ward in-patient / referred from A&E or another speciality) At least one ovarian cyst (excluding a corpus luteum)

Exclusion Criteria:

- Age <16 (so as to avoid problems with consent / Gillick competence) Not pregnant (ie. attending the unit with acute gynaecology problem or for follow up after a miscarriage) Lacks capacity to consent Corpus luteal cyst only on ultrasound scan

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women (diagnosed on urinary HCG) who attend the Early Pregnancy Unit at St. Thomas' Hospital and undergo an early pregnancy ultrasound scan. If the scan also shows one or more ovarian cysts, they are eligible for the study, as per the criteria above.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of ovarian cysts that are still visible at the final scan (6 weeks post partum) | 10 months

SECONDARY OUTCOMES:
The nature of the ovarian cysts (i.e functional/dermoid/endometrioma/borderline/malignant) | 10 months
The proportion of patients who required other imaging as well as ultrasound scans (eg. MRI) | 10 months
The prevalence of ovarian cysts in pregnancy | 16 months
The proportion of pregnant women who still have a corpus luteum at 20 weeks | 5 months
The proportion of pregnant woman with ovarian cysts who require surgical intervention | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Magee, MBChB, Principal Investigator — Guys and St. Thomas' NHS Foundatiuon Trust

IPD SHARING:
Plan to Share IPD: Undecided